CLINICAL TRIAL: NCT05209477
Title: Effects of Body Position and Recruiting Maneuver on Lung Aeration Assessed Through Ultrasound in Patients Intubated for Acute Respiratory Failure Related to Novel Coronavirus 19 Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera di Perugia (Other)
Responsible Party: Principal Investigator, Prof Gianmaria Cammarota, Prof Gianmaria Cammarota md, phd, Azienda Ospedaliera di Perugia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12/21
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung ultrasound (Other): n patients undergoing invasive mechanical ventilation with an arterial oxygen tension on inspired oxygen fraction ratio < 200 mmHg requiring recruitment maneuver and prone positioning as a rescue therapy, lung aeration will be evaluated at:
  baseline, in supine position under protective ventilation after two minute of recruitment maneuver in pressure controlled ventilation at 1 hour following prone positioning application
  Interventions: Other: lung ultrasound assessment

INTERVENTIONS:
Other: lung ultrasound assessment — In patients undergoing invasive mechanical ventilation with an arterial oxygen tension on inspired oxygen fraction ratio < 200 mmHg requiring recruitment maneuver and prone positioning as a rescue therapy, lung aeration will be evaluated at:
  1. baseline, in supine position under protective ventilation
  2. after two minute of recruitment maneuver in pressure controlled ventilation
  3. at 1 hour following prone positioning application

SUMMARY:
Second analysis of data prospectively collected during an investigation assessing the clinical characteristics of patients admitted for hypoxemic acute respiratory failure (hARF) related to novel coronavirus 19 disease (COVID-19). In particular, the primary aim of the present analysis is to assess the effects of recruiting maneuver and prone positioning on lung aeration evaluated through lung ultrasound in patients undergoing invasive mechanical ventilation

ELIGIBILITY:
Inclusion Criteria: Patients intubated for COVID-19 hARF -

Exclusion Criteria: Any contraindication to recruitment and lung ultrasound, pregnancy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
lung ultrasound score | after 20 minutes following study entry, in volume controll ventilation and supine position
  lung aeration evaluated through ultrasound during protective invasive mechanical in supine position. Lung ultrasound score ranges from a minimum of 0 to a maximum of 36, where 0 is the best lung aeration and 36 is the worst lung aeration
lung ultrasound score recruitment | 2 minutes
  lung aeration evaluated through ultrasound during protective invasive mechanical ventilation in supine position after two minutes of recruiting maneuver in pressure controlled ventilation. Lung ultrasound score ranges from a minimum of 0 to a maximum of 36, where 0 is the best lung aeration and 36 is the worst lung aeration
lung ultrasound score prone positioning | 1 hour
  lung aeration evaluated through ultrasound during protective invasive mechanical ventilation after 1 h from prone position application. Lung ultrasound score ranges from a minimum of 0 to a maximum of 36, where 0 is the best lung aeration and 36 is the worst lung aeration

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Perugia, Perugia, Umbria, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided